CLINICAL TRIAL: NCT06391463
Title: Analysis of the Presence of Multi-resistant and Spore-forming Bacteria in a Neonatal Intensive Care Unit: Implications for Practice
Brief Title: Multi-resistant and Spore-forming Bacteria in a Neonatal Intensive Care Unit
Acronym: NEOBIOTA
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5224
Record Dates: First submitted 2024-03-04; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Multidrug Resistant Bacterial Infection
Keywords: multidrug-resistant bacteria; neonatology; spore-forming bacteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infants admitted in the neonatal unit of croix rousse hospital: Infant born between January 1, 2018 and September 27, 2020, admitted in the neonatology department of the Croix Rousse hospital who had at least one coproculture during their stay
  Interventions: Other: Carriage of MRB ou BC

INTERVENTIONS:
Other: Carriage of MRB ou BC — Study of the epidemiology of the carriage of BMR and BC germs in patients in the neonatology department

SUMMARY:
Preventing the spread of multidrug-resistant bacteria (MRB) is a major challenge for hospitals today. MRB are defined as bacteria that combine several resistance mechanisms to different families of antibiotics, thus limiting therapeutic possibilities in the event of infection.

The spread of MRBs is particularly prevalent in hospital units caring for fragile patients, such as neonatal units. Preventing the spread of MRBs is of prime importance in these units, in order to limit the number of infections caused by these germs. Newborns are at risk of infection due to intrinsic factors such as an immature immune system and fragile skin, as well as extrinsic factors such as mechanical ventilation and intravascular catheters.

In Germany, a 2012 KRINKO agreement encourages neonatal units to monitor MRB carriage on a weekly basis. This measure enables early detection of MRB colonization outbreaks in neonatal units. In France, MRB carriage monitoring in neonatal units is not systematic.

Spore-forming bacteria also require close monitoring in neonatology, as they do not strictly meet the definition of MRB, but represent a major threat to newborns. The main spore-forming bacterium of medical interest is Bacillus cereus (BC), which is responsible for serious infections in premature infants. BC is resistant to the use of hydro-alcoholic solutions. The origin of these BC infections remains controversial, with numerous studies in the international literature suggesting a link between BC infections and contamination of breast milk given to infants in neonatal units. The role of environmental contamination has also been studied. The potential seriousness of these BC infections justifies the systematic detection of the carriage of this spore-forming bacterium in routine coprocultures, in the same way as other MRB germs.

In the neonatal unit at Hôpital de la Croix Rousse, MRB and BC are routinely tested on patient arrival, and then weekly until discharge.

If MRB or BC germs are found in children's stools reinforced specific hygiene measures are implemented to prevent cross-transmission in this open-bay unit with little space between incubators. Reinforced specific hygiene measures represent a time constraint for the nursing team, for parents and a financial burden for the neonatal unit. However, to our knowledge, there are no international or national recommendations concerning the duration of stools reinforced specific hygiene measures. Our clinical experience has shown that the persistence of pathogenic germs in stools seems to vary in duration depending on the microorganism.

To better determine the optimal duration of reinforced specific hygiene measures, as it is costly in terms of work time, parental stress, and hospital expenses due to reinforced hygiene conditions during the isolation period.

ELIGIBILITY:
* Inclusion Criteria * :

  * Children hospitalized in the department of neonatology at croix rousse university hospital
  * With at least one coproculture
* Exclusion Criteria * :

  * Death or discharge of the patient before the first stool culture has been taken
  * Impossibility for the laboratory to interpret the stool culture in a patient in whom only one stool culture has been taken, or recurrence of impossibility to interpret all stool cultures from the same patient.

Max Age: 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn hospitalized in the neonatology service of Croix Rousse hospital with at least one coproculture
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine the number of patients carrying BMR and BC germs | up to 4 months postnatal age or discharge which comes first
  Determine the number of patients carrying BMR and BC germs

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Croix Rousse, Lyon, France